CLINICAL TRIAL: NCT02325882
Title: The Postoperative Analgesic Effect of Combination With Dexmedetomidine in Fentanyl-based Intravenous Patient Controlled Analgesia Compared With Conventional Thoracic Epidural and Intravenous Patient Controlled Analgesia After Radical Open Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2014-0883
Record Dates: First submitted 2014-12-21; First posted 2014-12-25 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; 3-methylfentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conventional fentanyl-based epidural PCA (Active Comparator)
  Interventions: Drug: Fentanyl 1
- dexmedetomidine to fentanyl-based intravenous PCA (Experimental)
  Interventions: Drug: Dexmedetomidine
- Conventional fentanyl-based intravenous PCA (Active Comparator)
  Interventions: Drug: Fentanyl 2

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine mixed fentanyl based intravenous PCA
  Arms: dexmedetomidine to fentanyl-based intravenous PCA
Drug: Fentanyl 1 — conventional fentanyl-based epidural PCA
  Arms: Conventional fentanyl-based epidural PCA
Drug: Fentanyl 2 — conventional fentanyl based intravenous PCA
  Arms: Conventional fentanyl-based intravenous PCA

SUMMARY:
The aim of this study to test hypothesis that addition of dexmedetomidine to fentanyl based intravenous patient controlled analgesia (PCA) improves postoperative pain compared with conventional thoracic epidural and intravenous patient controlled analgesia after radical open gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. ASA class I-II
2. obtaining written informed consent from the parents
3. aged 20-65 years who were undergoing radical open gastrectomy

Exclusion Criteria:

1. abdominal surgery previously
2. patient who refuse the patient controlled analgesia
3. unstable angina or congestive heart failure
4. uncontrolled hypertension (diastolic bp>110mmHg)
5. coagulopathy
6. hepatic failure
7. renal failure
8. bradycardia on EKG (under 50 bpm)
9. Ventricular conduction abnormality
10. drug hyperactivity
11. neurological or psychiatric illnesses
12. mental retardation
13. patients who can't read the consent form due to illiterate or foreigner 14.infection

15. pregnant 16. obesity (BMI > 30kg/m2)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 48 hours after operation
  Postoperative pain measure using verbal numerical rating scales (VNRS) for 48 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, Seoul, South Korea